CLINICAL TRIAL: NCT01555086
Title: Prospective Randomized Study to Compare a Limited Versus Extended Pelvic Lymphadenectomy During Prostatectomy
Brief Title: Prospective Study to Compare a Limited Versus Extended Pelvic Lymphadenectomy During Prostatectomy
Acronym: SEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association of Urologic Oncology (AUO) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 55/09; DRKS00003256 (Registry Identifier: DRKS)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Lymphadenectomy; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Limited pelvic Lymphadenectomy (Experimental)
  Interventions: Procedure: Limited pelvic Lymphadenectomy
- Extended pelvic Lymphadenectomy (Experimental)
  Interventions: Procedure: Extended pelvic Lymphadenectomy

INTERVENTIONS:
Procedure: Limited pelvic Lymphadenectomy — approximately 10-14 lymph nodes are removed
  Other Names: limited pelvic LA
  Arms: Limited pelvic Lymphadenectomy
Procedure: Extended pelvic Lymphadenectomy — approximately 20 lymph nodes are removed
  Other Names: extended pelvic LA
  Arms: Extended pelvic Lymphadenectomy

SUMMARY:
This study examines Limited versus extended pelvic lymphadenectomy.

DETAILED DESCRIPTION:
This study is meant to show if the extension of lymphadenectomy during prostatectomy has an influence of outcome of patients. Patients with indication to prostatectomy due to prostate cancer will be included.

Both extensions of lymphadenectomy are used in hospitals as a free choice. This study shell show if one method is more effective than the other.

ELIGIBILITY:
Inclusion Criteria:

* stamp bioptic secured prostate cancer with intermediate or high risk profile (defined as Gleason-Score 7-10 or PSA > 10 ng/ml)
* locally-operable tumor according to DRU/TRUS
* negative bone scan
* negative CT abdomen / pelvis
* general condition according to Karnofsky >/= 80%
* written consent of the patient
* adequate hematological, renal and coagulation physiological functions
* Patient compliance and geographic proximity to allow adequate follow-up

Exclusion Criteria:

* Manifest secondary malignancy
* Secured metastasis by histologically or by imaging
* Myocardial infarction or stroke within the last 6 months
* Existing major cardiovascular (grade III - IV according to NYHA), pulmonary (pO2 <60 mmHg), renal, hepatic or hematopoietic (eg severe bone marrow aplasia) diseases
* Severe active or chronic infections (eg pos. HIV-Ab test, HBs-Ag detection in serum and / or chronic hepatitis)
* severe psychiatric disease
* prior chemotherapy (allowed is a preoperative antiandrogen therapy ≤ 3 months)
* previous pelvic radiotherapy
* Patients in a closed institution according to an authority or court decision
* People who are in a dependent relationship or working relationship with the sponsor or investigator
* simultaneous participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
PSA-progress | 5 years
  3-monthly Follow-up with PSA-measurement in blood

SECONDARY OUTCOMES:
Comparison of overall survival | 5 years
  Comparison of overall survival after limited versus extended lymphadenectomy after prostatectomy
Comparison of morbidity | 5 years
  Comparison of morbidity after limited versus extended lymphadenectomy after prostatectomy

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Krankenhaus Maria Hilf, Krefeld, Dießemer Bruch 80
  - Martiniklinik am UKE, Hamburg, Martinistraße 52
  - St. Antonius-Krankenhaus, Gronau, Möllenweg 22
  - Städtisches Klinikum Fulda, Fulda, Pacelliallee 3-5
  - RWTH Aachen, Aachen, Pauwelsstraße 30